CLINICAL TRIAL: NCT00195923
Title: Prospective Randomized Evaluation of Antibiotic Regimen Following Appendectomy for Perforated Appendicitis
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: 04-12-149
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2005-09

CONDITIONS: Perforated Appendicitis
Keywords: appendicitis; perforation
MeSH Terms: conditions — Appendicitis | interventions — Ampicillin; Gentamicins; Clindamycin; Metronidazole; Ceftazidime

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ampicillin, gentamicin, clindamycin, flagyl, ceftazidime

SUMMARY:
The purpose of this study is to compare traditional triple antibiotic therapy against dual single day dosing antibiotic therapy in the management of perforated appendicitis in children.

DETAILED DESCRIPTION:
Triple antibiotic therapy providing broad spectrum coverage of gram positive, gram negative and anaerobic bacteria has long been the standard treatment for perforated appendicitis in children. This regimen has traditionally consisted of ampicillin, gentamicin, and clindamycin. The dosing regimen for these medications are quite frequent, as follows: ampicillin (every 6 hours), gentamicin (every 8 hours), and clindamycin (every 8 hours), until there is no evidence for postoperative infection, usually 5 to 7 days. Further, gentamicin is an aminoglycoside with known renal and ototoxic side effects. Its therapeutic window is small necessitating measurement of serum levels to maintain therapeutic levels and avoid toxicity. The contemporary selection of antibiotics includes very few drugs that require such monitoring.

Monotherapy with newer broad-spectrum agents such as piperacillin/tazobactam for intraabdominal infections has recently been demonstrated to be equally efficacious as traditional triple therapy. Such data calls into question the need for such onerous antibiotic regimens which include a nephrotoxic agent (gentamycin). However, the benefits of monotherapy are outweighed by the increased expense of the antibiotic, and the ongoing cumbersome dosing schedule of 3-4 doses daily. We have recently moved to a dual antibiotic regimen (ceftriaxone and metronidazole) which provides excellent antimicrobial coverage and can be dosed on a once daily dosing schedule with an identical duration of therapy as for the triple antibiotic regimen. This regimen has proven effective in adults with intraabdominal infections such as perforated appendicitis. Further, ceftriaxone plus metronidazole has been shown equal to the aforementioned monotherapy schedule with piperacillin/tazobactam in children with complicated perforated appendicitis. The advantages of dual antibiotic therapy with once a day dosing for children with perforated appendicitis are immense, especially if the antibiotics are well tolerated, less expensive, and have a simple dosing schedule. Additionally, neither drug is nephrotoxic; both have broad therapeutic ranges and therefore require no serum level measurements. This translates into less blood draws, less time patients need to be receiving infusions, and less utilization of nursing resources. These advantages would be expected to culminate in greater nursing and patient satisfaction. The purpose of this study is to scientifically compare the traditional triple antibiotic regimen to dual antibiotic regimen for children with perforated appendicitis, quantify its significance, and report our findings to physicians caring for these children.

This will be a prospective randomized study involving children who undergo appendectomy for perforated appendicitis. All patients will receive antibiotics (ceftriaxone and flagyl) preoperatively. The determination of perforation will be made by the surgeon at the time of the operation. Perforation will be determined by either identifying a perforation in the appendix itself, or by identifying anaerobic odors emanating from the abdominal cavity during operation (sniff test). Once perforated appendicitis has been documented, the parents/guardians of the patient will be informed of the option to participate in the prospective randomized study. Patients whose parents agree and consent to enroll in the study will then be randomized to one of 2 groups based on a sequential randomization number created by Steve Simon, PhD.

Based on a power analysis of length of stay, performed by Dr. Simon, 50 patients in each of the two arms of the study will provide a power of 82% with an alpha level of 0.05. Dr. Simon feels that this level is appropriate for this study.

The control group will consist of triple antibiotic coverage with ampicillin 50mg/kg every 6 hours, gentamicin 2.5 mg/kg every 8 hours and clindamycin 10mg/kg every 6 hours, which are standard dosing regimens. The experimental group will receive ceftriaxone 50mg/kg once a day (maximum dose = 2 grams) and metronidazole 30mg/kg once a day (maximum dose = 1 gram) with once a day dosing for both. The length of antibiotic therapy will not differ from our standard management and will remain standardized in both arms. All patients will receive a minimum of 5 days of therapy (regardless of group randomization). At that time, if they have been afebrile for at least 24 hours, a white blood cell (WBC) count will be obtained, and if that is within normal limits, the antibiotics will be discontinued. If, after 5 days of therapy, the patient remains febrile, therapy will continue without change, unless cultures obtained from the febrile response indicate a need for antibiotic coverage change. If a change in antibiotic regimen is indicated, the antibiotic profile will be evaluated and the most appropriate antibiotic will be instituted. If this occurs, the patient's data will continue to be collected in an intention to treat analysis. In cases where there is no indication for a change in antibiotic regimen, a WBC count will be drawn once the patient has become and remains afebrile for a complete 24 hour period of time. If the WBC is elevated, the antibiotic course will continue with WBC counts to be drawn daily until normal values return. If leukocytosis or fever persists for 10 days, or if there is clinical indication of a postoperative intra-abdominal infection, a CT scan of the abdomen and pelvis will be performed to determine if a postoperative abscess has developed. Identification of a postoperative abscess will result in percutaneous drainage with culture and sensitivity of the abscess fluid. Subsequent antibiotic treatment will be based on the sensitivities obtained from the culture of the abscess. In these cases the patients' data will be collected and they will be regarded as a failure of antibiotic therapy in the final analysis.

Parental permission and child assent, if the child is old enough, will be obtained (see attached form) and patients will be randomized to the control or experimental group based on a randomization number generated by Dr. Steve Simon, PhD. Patient demographics, operative approach, time to tolerating full feeds, length of hospitalization, infectious complications, medication charges, and hospital charges will be collected for comparison between the groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients under 18 years of age found to have perforated appendicitis at the time of operation for appendicitis and whose parents give informed permission will be included in the study.

Exclusion Criteria:

* Patients with a normal or non-perforated appendix at the time of appendectomy, those without parental permission, or those with a documented allergy to any of the antibiotics used in either regimen will be excluded from the study. Patients 18 years or older will not be included in the study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2005-04; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Ostlie, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States